CLINICAL TRIAL: NCT03551002
Title: Impact of Direct Acting Antivirals Uptake in Controlling Hepatitis C Epidemic and Modeling Interventions for Hepatitis C Elimination Among HIV-infected Persons in San Diego
Brief Title: Impact of DAA Uptake in Controlling HCV Epidemic and Modeling Interventions for HCV Elimination Among HIV-infected Persons in San Diego
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Cachay, MD, MAS, Associate Professor of Clinical Medicine, University of California, San Diego
Other Study IDs: IN-US-334-4481; 171954 (Other: UCSD Human Research Protections Program)
Record Dates: First submitted 2018-05-23; First posted 2018-06-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C; Hepatitis C, Chronic; HIV/AIDS
Keywords: HIV; Hepatitis C; Direct acting antivirals; Hepatitis C modeling
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — For patients who fail direct acting antivirals (DAA) therapy, a blood sample will be collected to conduct phylogenetic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective
- Prospective

SUMMARY:
A retrospective and prospective study among people living with HIV (PLWH) that assesses hepatitis C (HCV) treatment uptake during periods before and after direct acting antivirals (DAA) introduction, and its impact on the HCV epidemic among PLWH.

DETAILED DESCRIPTION:
A study that aims to quantify the state of DAA uptake and its impact on the HCV epidemic among PLWH in San Diego, and to characterize negative predictors of DAA treatment uptake among PLWH in San Diego. Retrospective and prospective data from UCSD Owen Clinic will be utilized to calculate HCV prevalence, primary incidence, and reinfection incidence. Using mathematical epidemic models, the study will assess levels of existing and scaled-up interventions necessary for HCV elimination from PLWH in San Diego.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 years) HIV-infected patient attending the UCSD Owen Clinic
* With history of acute or chronic HCV infection defined as having a detectable HCV viral load with or without a positive HCV antibody

Exclusion Criteria:

* With no history of or current HCV infection defined as having a negative HCV antibody from 2008 to 2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV, with history of or current HCV infection, who receive care at the UCSD Owen Clinic from 2008 to 2020
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual proportion of HIV-infected patients who initiate direct acting antivirals | 2014-2020

SECONDARY OUTCOMES:
Annual proportion of PLWH co-infected with HCV who are treatment naïve, previously treated with no sustained virologic response (SVR), or re-infected post-SVR | 2008-2020
Annual HCV chronic prevalence, primary incidence, and reinfection incidence among HIV-infected patients | 2008-2020

OTHER OUTCOMES:
Estimated HCV prevalence and incidence among PLWH in San Diego using dynamic transmission modeling calibrated to epidemiological data from outcomes described above | 2008-2030

CONTACTS AND LOCATIONS:
Overall Officials: Edward Cachay, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- Owen Clinic-University of California, San Diego, San Diego, California, United States